CLINICAL TRIAL: NCT01656642
Title: A Phase Ib, Open-Label Study of The Safety and Pharmacology of Atezolizumab (Anti PD-L1 Antibody) Administered in Combination With Vemurafenib or Vemurafenib Plus Cobimetinib in Patients With BRAFV600-Mutation Positive Metastatic Melanoma
Brief Title: A Phase 1b Study of Atezolizumab in Combination With Vemurafenib or Vemurafenib Plus Cobimetinib in Participants With BRAFV600-Mutation Positive Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GP28384; 2012-002738-35 (EudraCT Number)
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Malignant Melanoma
Keywords: PD-L1; PD-1; PDL1; antiPD-L1; MPDL3280A; Melanoma; BRAF; MPDL320A
MeSH Terms: conditions — Melanoma | interventions — atezolizumab; cobimetinib; Vemurafenib

ARMS (7):
- Cohort 1 (C1): Ate+Vem - No Run-in (Experimental): Participants will receive atezolizumab (Ate) 1200 milligrams (mg) every 3 weeks (q3w) along with vemurafenib (Vem) 720 mg twice daily (BID) for 21 days in each cycle followed by 7 days off treatment (28-day cycle). Treatment will continue until disease progression, unacceptable toxicity, or withdrawal of consent occurs.
  Interventions: Drug: Atezolizumab; Drug: Vemurafenib
- Cohort 2 (C2): Ate+Vem (56 Day Run-in) (Experimental): Run-in period (56 days): participants will receive vemurafenib 960 mg orally BID from Day 1 to 49 and vemurafenib 720 mg orally BID from Day 50 to 56. Combination treatment period: Participants will receive fixed dose of atezolizumab 1200 mg intravenous (IV) q3w in combination with vemurafenib 720 mg orally BID in 21 days cycle.
  Interventions: Drug: Atezolizumab; Drug: Vemurafenib
- Cohort 3 (C3): Ate+Vem (28 Day Run-in) (Experimental): Run-in period (28 days): participants will receive vemurafenib 960 mg orally BID for 21 days, then vemurafenib 720 mg orally BID for 7 days. Combination treatment period: Participants will receive fixed dose of atezolizumab 1200 mg IV q3w in combination with vemurafenib 720 mg orally BID in 21 days cycle.
  Interventions: Drug: Atezolizumab; Drug: Vemurafenib
- Cohort 4 (C4): Ate+Vem+Cob (28 Day Run-in) (Experimental): Run-in period (28 days): participants will receive vemurafenib 960 mg orally BID for 21 days, then vemurafenib 720 mg orally BID for 7 days in combination with cobimetinib (Cob) 60 mg IV once daily, 21 days on/7 days off schedule (21/7). Combination treatment period: Participants will receive fixed dose of atezolizumab 800 mg IV every 2 weeks (q2w) in combination with vemurafenib 720 mg orally BID and cobimetinib 60 mg orally once daily 21/7 in 28 days cycle.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib; Drug: Vemurafenib
- ECA: Ate+Vem+Cob (Mandatory Biopsy PD) (Experimental): Expansion Cohort A (ECA): Approximately 10 participants who experienced disease progression (PD) after receiving prior checkpoint inhibitor therapy will be enrolled and treated with atezolizumab plus (+) vemurafenib + cobimetinib. Serial biopsy tissue sample collections of accessible lesions will be mandatory for all participants enrolled in this cohort. The doses will be decided based on the results of Cohorts 1-4.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib; Drug: Vemurafenib
- ECB: Ate+Vem+Cob (Mandatory Biopsy) (Experimental): Expansion Cohort B (ECB): Approximately 20 participants will be enrolled and treated with atezolizumab + vemurafenib + cobimetinib. Serial biopsy tissue sample collections of accessible lesions will be mandatory for all participants. The doses will be decided based on the results of Cohorts 1-4.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib; Drug: Vemurafenib
- ECC: Ate+Vem+Cob (No Mandatory Biopsy) (Experimental): Expansion Cohort C (ECC): Approximately 10 participants who experienced disease progression after receiving prior checkpoint inhibitor therapy will be enrolled and treated with atezolizumab + vemurafenib + cobimetinib. Serial biopsy tissue sample collections will be optional for all participants enrolled in this cohort. The doses will be decided based on the results of Cohorts 1-4.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib; Drug: Vemurafenib

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered q3w or q2w.
  Other Names: MPDL3280A, an engineered anti-PD-L1 antibody; TECENTRIQ; RO5541267
Drug: Cobimetinib — Oral repeating dose
  Other Names: GDC-0973; XL518; Cotellic; RO5514041
  Arms: Cohort 4 (C4): Ate+Vem+Cob (28 Day Run-in); ECA: Ate+Vem+Cob (Mandatory Biopsy PD); ECB: Ate+Vem+Cob (Mandatory Biopsy); ECC: Ate+Vem+Cob (No Mandatory Biopsy)
Drug: Vemurafenib — Oral repeating dose, depending on arm/cohort
  Other Names: Zelboraf; RO5185426

SUMMARY:
This is an open-label, multicenter, Phase Ib, dose-escalation and cohort-expansion study of atezolizumab (anti-programmed death-ligand 1 [PD-L1] antibody) in combination with vemurafenib or vemurafenib plus cobimetinib in participants with BRAFV600-mutation positive metastatic melanoma. Enrolled participants may continue treatment until they are no longer experiencing clinical benefit as assessed by the investigator and in alignment with the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic documentation of metastatic or Stage IIIc unresectable melanoma, with BRAFV600 mutation as assessed by BRAFV600 Mutation Test. Origin of the primary tumor may be of skin, mucosal, or acral locations but not of uveal origin. Participants having an unknown primary tumor may be eligible if uveal melanoma can be ruled out
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Adequate hematologic and end organ function
* Measurable disease per RECIST v1.1
* For women of childbearing potential, agreement to remain abstinent (refrain from heterosexual intercourse) or use two effective forms of contraceptive methods including at least one that results in a failure rate of less than (<) 1 percent (%) per year during the treatment period and for at least 6 months after the last dose of study drug
* For men, agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm
* Agreement to mandatory archival tissue or fresh biopsy
* Agreement to the collection of serial fresh lesion samples (required, if feasible, for entry into Escalation Cohorts 4 and Expansion Cohorts A & B and optional, but encouraged in Escalation Cohorts 2 & 3 and Expansion Cohort C)

Exclusion Criteria:

* Receipt of prior systemic anti-cancer therapy for unresectable, locally advanced or metastatic melanoma
* Receipt of prior immunomodulatory agents, including programmed death-1 or PD-L1 targeted therapy or cytotoxic T-lymphocyte-associated antigen 4 targeted therapy including ipilimumab (this exclusion criterion does not apply to participants enrolled in Expansion Cohort A)
* Receipt of prior mitogen-activated protein kinase inhibitor pathway agents including mitogen-activated protein kinase inhibitor and BRAF kinase inhibitor
* Major surgical procedure within 28 days prior to Day 1 or anticipation of need for a major surgical procedure during the course of the study
* Radiotherapy less than or equal to (<=) 7 days prior to Day 1
* Adverse events from prior anti-cancer therapy that have not resolved to Grade <= 1 except for alopecia
* Any active malignancy (other than BRAF-mutated melanoma) or a previous malignancy within the past 3 years
* For participants to be enrolled into the vemurafenib+cobimetinib+ atezolizumab cohorts: history of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment/central serous chorioretinopathy, retinal vein occlusion, or neovascular macular degeneration
* Pregnant or breastfeeding women
* Intake of St. John's wort or hyperforin (potent cytochrome P450 [CYP] 3A4 enzyme inducer) or grapefruit juice (potent CYP3A4 enzyme inhibitor) within 7 days preceding the start of study treatment to the end of treatment
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation or known hypersensitivity to any component of cobimetinib or vemurafenib
* Inability to comply with study and follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-08-13 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose Limiting Toxicities | 21 days (or 28 days for Cohort 4) following the first administration of atezolizumab
Percentage of Participants With Adverse Events | Baseline up to approximately 6 years

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC) of Atezolizumab | Predose (0 hour), 30 minutes postdose on Day (D) 1 of Cycles (C) 1, 2; predose on D15, D8 of C1; predose on D1 of C3, 4, 5, 7, 8, every 8 cycles thereafter up to 90 days after end of treatment visit (up to approximately 6 years) (Cycle=28 days)
Maximum Serum Concentration of Atezolizumab | Predose (0 hour), 30 minutes postdose on Day (D) 1 of Cycles (C) 1, 2; predose on D15, D8 of C1; predose on D1 of C3, 4, 5, 7, 8, every 8 cycles thereafter up to 90 days after end of treatment visit (up to approximately 6 years) (Cycle=28 days)
Maximum Plasma Concentration of Vemurafenib | Run-in period: predose (0 hour) on D1, 8, and 22, 3 hours postdose on D22; combination treatment period: predose (0 hour) on D1 of C1 and 2, 3 hours postdose on D1 of C2 (Cycle = 28 days)
Minimum Observed Plasma Trough Concentration (Cmin) of Vemurafenib | Run-in period: predose (0 hour) on D1, 8, and 22; combination treatment period: predose (0 hour) on D1 of C1 and 2 (Cycle = 28 days)
Maximum Plasma Concentration of Cobimetinib | Run-in period: predose (0 hour) on D1, 8, and 22; combination treatment period: predose (0 hour) on D1 and 15 of C1 and D15 of C2, 3 hours postdose on D15 of Cycle 1 (Cycle = 28 days)
Cmin of Cobimetinib | Run-in period: predose (0 hour) on D1, 8, and 22; combination treatment period: predose (0 hour) on D1 and 15 of C1 and D15 of C2 (Cycle = 28 days)
Percentage of Participants With Best Overall Response According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1) | Baseline until disease progression or death, whichever occurred first (assessed at baseline, every 6 weeks of combination treatment period for first 24 weeks and then every 9 weeks up to approximately 6 years)
Percentage of Participants with Objective Response According to RECIST v1.1 | Baseline until disease progression or death, whichever occurred first (assessed at baseline, every 6 weeks of combination treatment period for first 24 weeks and then every 9 weeks up to approximately 6 years)
Percentage of Participants with Objective Response According to Immune-Related Response Criteria (irRC) | Baseline until disease progression or death, whichever occurred first (assessed at baseline, every 6 weeks of combination treatment period for first 24 weeks and then every 9 weeks up to approximately 6 years)
Duration of Objective Response According to RECIST v1.1 | Baseline until disease progression or death, whichever occurred first (assessed at baseline, every 6 weeks of combination treatment period for first 24 weeks and then every 9 weeks up to approximately 6 years)
Duration of Objective Response According to irRC | Baseline until disease progression or death, whichever occurred first (assessed at baseline, every 6 weeks of combination treatment period for first 24 weeks and then every 9 weeks up to approximately 6 years)
Progression Free Survival According to RECIST v1.1 | Baseline until disease progression or death, whichever occurred first (assessed at baseline, every 6 weeks of combination treatment period for first 24 weeks and then every 9 weeks up to approximately 6 years)
Progression Free Survival According to irRC | Baseline until disease progression or death, whichever occurred first (assessed at baseline, every 6 weeks of combination treatment period for first 24 weeks and then every 9 weeks up to approximately 6 years)
Overall Survival Duration | Baseline until death up to 6 years
Mean Atezolizumab Dose | Approximately 12 months
Total Number of Atezolizumab Cycles | Approximately 12 months
Percentage of Participants With Anti-Atezolizumab Antibodies | Predose (0 hour) on D1 (run-in period), predose (0 hour) on D1 of C2, 3, 4, 8, every 8 cycles thereafter up to 90 days after end of treatment visit (up to approximately 6 years) (Cycle=28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (8):
- United States (8):
  - UCLA, Los Angeles, California
  - The Angeles Clinic and Research Institute - W LA Office, Los Angeles, California
  - University of Colorado Health Science Center; Biomedical Research Bldg. Room 511, Aurora, Colorado
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Massachusetts General Hospital., Boston, Massachusetts
  - Dana Farber Can Ins, Boston, Massachusetts
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Sullivan RJ, Hamid O, Gonzalez R, Infante JR, Patel MR, Hodi FS, Lewis KD, Tawbi HA, Hernandez G, Wongchenko MJ, Chang Y, Roberts L, Ballinger M, Yan Y, Cha E, Hwu P. Atezolizumab plus cobimetinib and vemurafenib in BRAF-mutated melanoma patients. Nat Med. 2019 Jun;25(6):929-935. doi: 10.1038/s41591-019-0474-7. Epub 2019 Jun 6. PMID 31171876
- [Derived] Ackerman A, Klein O, McDermott DF, Wang W, Ibrahim N, Lawrence DP, Gunturi A, Flaherty KT, Hodi FS, Kefford R, Menzies AM, Atkins MB, Long GV, Sullivan RJ. Outcomes of patients with metastatic melanoma treated with immunotherapy prior to or after BRAF inhibitors. Cancer. 2014 Jun 1;120(11):1695-701. doi: 10.1002/cncr.28620. Epub 2014 Feb 27. PMID 24577748